CLINICAL TRIAL: NCT04118491
Title: Hyperbaric Oxygen for Carbon Monoxide Induced Chronic Encephalopathy
Acronym: HACMICE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 0225-18-FB
Record Dates: First submitted 2019-07-26; First posted 2019-10-08 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Carbon Monoxide Poisoning; Chronic Encephalopathy
MeSH Terms: conditions — Carbon Monoxide Poisoning; Brain Damage, Chronic

STUDY DESIGN:
Intervention Model Description: treating with hyperbaric oxygen therapy vs sham in a randomized crossover fashion
Who Masked: Participant
Masking Description: sham control- sham HBO2 treatments (air at near normal pressure (1.2 ATA)). Treatments will be done once daily for 2 hours, Monday through Friday.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- sham1st (Sham Comparator): 40 sham HBO2 treatments (air at near normal pressure (1.2 ATA)). Treatments will be done once daily for 2 hours, Monday through Friday. The second block will be treated similarly except that they will receive sham treatments in the first block and oxygen treatments in the second block.
  Interventions: Device: hyperbaric oxygen and sham hyperbaric oxygen
- sham second (Active Comparator): iii. We will divide the subjects into two groups of five. One group will receive 40 Hyperbaric Oxygen (HBO2) treatments (100% oxygen at twice normal air pressure (2 ATA)) followed by 40 sham HBO2 treatments (air at near normal pressure (1.2 ATA)). Treatments will be done once daily for 2 hours, Monday through Friday. The second block will be treated similarly except that they will receive sham treatments in the first block and oxygen treatments in the second block.
  iv. Neurological and psychologic assessments will be done prior to starting treatments, after the first block of 40 and again after the second block of 40.
  Interventions: Device: hyperbaric oxygen and sham hyperbaric oxygen

INTERVENTIONS:
Device: hyperbaric oxygen and sham hyperbaric oxygen — see arm descriptions

SUMMARY:
In some patients, a few days or weeks after recovery from carbon monoxide poisoning, new symptoms develop. These can affect mood, ability to think or remember clearly, and movements. Some people develop movement problems that are similar to Parkinson's disease. This damage to brain tissue is called "encephalopathy," and this study will look at the effect of pressurized oxygen therapy on long term, or chronic, encephalopathy.

DETAILED DESCRIPTION:
Carbon monoxide (CO) poisoning is a leading cause of unintentional poisoning deaths in the United States. After a period of apparent recovery, survivors of acute CO-poisoning can develop a potentially permanent neurologic deterioration (DNS). DNS is a rare, poorly known encephalopathy with a 25-50% prevalence among severely poisoned CO-poisoned patients. Its symptoms and signs range from subtle abnormalities to severe dementia, Parkinsonism, gait disturbances, mutism, and incontinence. Recovery from delayed neuropsychiatric syndrome occurs in 50-75% of patients within 1 year. However, this leaves 25-50% permanently impaired.

Hyperbaric oxygen therapy (HBO2) is useful after acute poisoning to reduce the chance of developing DNS. However, appropriate therapy for DNS is widely debated; particularly, the role of hyperbaric oxygen therapy (HBO2) after DNS has developed is controversial. This study proposes to ascertain whether hyperbaric oxygen is efficacious in the treatment of chronic DNS brain injury from carbon monoxide (CO) poisoning. Ten participants suffering from DNS for longer than one year will be recruited to the study, which will be prospective, blinded, sham-controlled and crossover in design. Participants will be divided into two groups of five. One group will receive 40 HBO2 treatments [100% oxygen at twice normal air pressure (2 ATA)] followed by 40 sham HBO2 treatments [air at near normal pressure (1.2 ATA)]. Treatments will be done once daily for 2 hours, Monday through Friday. Neurological and psychologic assessments will be done prior to starting treatments, after each group of 40 treatments. The second group will be treated similarly except that they will receive sham treatments in the first and oxygen treatments second. In this manner, all participants will act as both experimental and control subject and will receive treatment which we believe is therapeutic.

ELIGIBILITY:
Inclusion Criteria:

* CO induced neurological or cognitive sequelae assessed as at least mild (e.g. UPDRS part 3 (motor)>15).
* chronicity- signs or symptoms present for greater than one year after exposure.

Exclusion Criteria:

* age >90 or less than 10 years
* other morbidities which may contribute to chronic neurocognitive deficits (such as traumatic brain injury, poisoning by other toxins, other neurodegenerative diseases)
* pregnancy (if a subject becomes pregnant she will be removed from the study)
* routine contraindications to hyperbaric oxygen

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Short Form (36) Health Survey | 4 months (after 80 treatments)
  is a 36-item, patient-reported survey of patient health

SECONDARY OUTCOMES:
Updrs part 3 (motor function) | 0, 2 and 4 months: (prior to study, after 40 treatments and 80 treatments)
  Unified Parkinson Disease Rating Scale
BARS- Brief Ataxia Rating Scale | 0, 2 and 4 months: (prior to study, after 40 treatments and 80 treatments)
  an assessment of ataxia, 30 point scale with 0 being normal
Fahn-Marsden Dystonia Rating Scale | 0, 2 and 4 months: (prior to study, after 40 treatments and 80 treatments)
  an assessment of dystonia, 120 point scale with 0 being normal
Physician assessment | prior to study, after 40 treatments and 80 treatments (0, 2 and 4 months)
  an assessment of global function, this is a verbal description not a scale
The Montreal Cognitive Assessment | 0, 2 and 4 months: (prior to study, after 40 treatments and 80 treatments)
  a brief cognitive screening tool for Mild Cognitive Impairment
Short Form (36) Health Survey | 0, 2 and 4 months: (prior to study, after 40 treatments and 80 treatments)
  is a 36-item, patient-reported survey of patient health

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Cooper, MD, Principal Investigator — University of Nebraska